CLINICAL TRIAL: NCT02157402
Title: A Youth Led Social Marketing Campaign to Encourage Healthy Lifestyles. EYTO (European Youth Tackling Obesity): A Randomized Controlled Trial in Catalonia (Spain)
Brief Title: EYTO (European Youth Tackling Obesity): A Randomized Controlled Trial in Catalonia (Spain)
Acronym: EYTO-SPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: European Commission (Other); Centro Tecnológico de Nutrición y Salud (Other); Hospital Universitari Sant Joan de Reus (Other); Companhia de Ideas (Unknown); Komunikujeme (Other); National Children's Bureau (Unknown)
Responsible Party: Principal Investigator, Rosa Sola, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EYTO-SPAIN
Record Dates: First submitted 2014-05-28; First posted 2014-06-06 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Life Style
Keywords: Adolescent
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The intervention group will received activities and social events designed according 8 social marketing Benchmark criteria to promote healthy lifestyles.
  Interventions: Behavioral: Social marketing activities and pop-up events to promote healthy lifestyles
- Control Group (No Intervention): The control group will not received any intervention activities and social events to promote healthy lifestyles.

INTERVENTIONS:
Behavioral: Social marketing activities and pop-up events to promote healthy lifestyles
  Arms: Intervention Group

SUMMARY:
Our hypothesis is that healthy lifestyles improvement by an intervention designed according 8 social marketing Benchmark criteria, can reduce overweight or obesity implemented by adolescents on their colleges.

The general aim of EYTO program is to improve health and well-being among adolescents who live in low socioeconomically communities, through an intervention study designed by selected adolescents with the inclusion of social marketing Benchmark criteria.

DETAILED DESCRIPTION:
5 adolescent coordinators (of intervention high-schools) will be trained by experts in social marketing and health promotion. This 5 selected adolescent as coordinators who will be in charge of the design of an 8 social marketing criteria intervention to implement their peers´ lifestyles.

The program has over two academic years. The participants will be followed for the duration of 2 academic years, an expected of up to 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by parents and/or guardians.
* Adolescents between 13 and 17 years old.

Exclusion Criteria:

- The lack of one or more inclusion criteria.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of Fruit intake | Change from Baseline in fruit Intake at 2 academic years
  Health Behaviour in School-aged Children (HBSC) survey
Change of Vegetable intake | Change from Baseline in vegetable Intake at 2 academic years
  Health Behaviour in School-aged Children (HBSC) survey
Change of Physical activity practice | Change from Baseline in physical activity practice at 2 academic years
  Health Behaviour in School-aged Children (HBSC) survey

SECONDARY OUTCOMES:
Change of Sedentary behaviour | Change from Baseline in sedentary behaviour at 2 academic years
  Health Behaviour in School-aged Children (HBSC) survey

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà Alberich, M.D., PhD, Principal Investigator — Centro Tecnológico de Nutrición y Salud
Locations (1):
- Universitat Rovira i Virgili, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Aceves-Martins M, Llaurado E, Tarro L, Papell-Garcia I, Prades-Tena J, Kettner-Hoeberg H, Puiggros F, Arola L, Davies A, Giralt M, Sola R. "Som la Pera," a School-Based, Peer-Led Social Marketing Intervention to Engage Spanish Adolescents in a Healthy Lifestyle: A Parallel-Cluster Randomized Controlled Study. Child Obes. 2022 Dec;18(8):556-571. doi: 10.1089/chi.2021.0207. Epub 2022 Mar 7. PMID 35255220
- [Derived] Llaurado E, Aceves-Martins M, Tarro L, Papell-Garcia I, Puiggros F, Arola L, Prades-Tena J, Montagut M, Moragas-Fernandez CM, Sola R, Giralt M. A youth-led social marketing intervention to encourage healthy lifestyles, the EYTO (European Youth Tackling Obesity) project: a cluster randomised controlled0 trial in Catalonia, Spain. BMC Public Health. 2015 Jul 3;15:607. doi: 10.1186/s12889-015-1920-1. PMID 26137843